CLINICAL TRIAL: NCT05631730
Title: An Investigator-Initiated Prospective Randomized Open-Label Blinded-Endpoint Crossover Trial Comparing the Effect and Safety of Flecainide and Metoprolol Versus Metoprolol Alone to Suppress Ventricular Arrhythmias in Arrhythmic Mitral Valve Prolapse
Brief Title: Effect and Safety of Flecainide and Metoprolol Versus Metoprolol Alone to Suppress Ventricular Arrhythmias in Arrhythmic Mitral Valve Prolapse
Acronym: FLECAPRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Eivind Westrum Aabel, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-500814-24-00; 2022-500814-24-00 (Other: European Union Clinical Trial Register)
Record Dates: First submitted 2022-11-08; First posted 2022-11-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mitral Valve Prolapse; Ventricular Arrhythmias and Cardiac Arrest
Keywords: arrhythmic mitral valve prolapse; mitral annular disjunction; ventricular arrhythmia
MeSH Terms: conditions — Mitral Valve Prolapse; Heart Arrest | interventions — Flecainide; Metoprolol

STUDY DESIGN:
Intervention Model Description: Crossover prospective randomized open-label blinded-endpoint (PROBE) trial.
Who Masked: Outcomes Assessor
Masking Description: Separate endpoint adjudication committee blinded to randomized allocation of patients to treatment groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flecainide and Metoprolol (Experimental): Participants will receive flecainide 50 mg twice daily (BID), with a dosage target of 100 mg BID. The maximum daily dose of flecainide will not exceed 300 mg. The first dose of flecainide will be initiated in-hospital with a 12-lead electrocardiogram (ECG) taken after 3 hours. If the ECG is considered normal after flecainide treatment, the participant will continue with 50 mg BID from the next day. Participants will receive a dosage of Metoprolol taking into consideration prior beta-blocker use and concomitant medications. The maximum daily dose of metoprolol will not exceed 200 mg. Within the run-in period, the dosage of both Flecainide and Metoprolol will be increased to the maximum tolerable dose.
  The Study Team can change the immediate-release formulation of Flecainide to controlled release at the same daily dose of flecainide. Whether metoprolol sustained release will be dosed once daily (QD) or BID, will be up to the investigator and patient preference.
  Interventions: Drug: Flecainide; Drug: Metoprolol
- Metoprolol Alone (Active Comparator): Participants will receive a dosage of Metoprolol taking into consideration prior beta-blocker use and concomitant medications. Within the run-in period, the dosage will be increased to the maximum tolerable dose. Whether metoprolol sustained release will be dosed QD or BID, will be up to the investigator and patient preference. The maximum daily dose of metoprolol will not exceed 200 mg.
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Flecainide — Flecainide is mainly used for pharmacological conversion in patients with atrial tachyarrhythmias and to suppress ventricular arrhythmias in patients with structurally normal hearts.
  Other Names: C01B C04
  Arms: Flecainide and Metoprolol
Drug: Metoprolol — Metoprolol is a beta-blocker and class II antiarrhythmic drug considered standard care in most cardiac diseases predisposing to ventricular arrhythmias, including arrhythmic mitral valve prolapse.
  Other Names: C07A B02

SUMMARY:
FLECAPRO is a randomized controlled crossover trial assessing the effect and safety of adding flecainide to standard beta-blocker therapy to reduce the burden of ventricular arrhythmias in patients with arrhythmic mitral valve prolapse. The primary endpoint of will be assessed using an implantable loop recorder with blinded endpoint adjudication.

DETAILED DESCRIPTION:
Mitral valve prolapse (MVP) is a common condition characterized by bulging one or both mitral leaflets into the left atrium. Although mainly a benign cardiac condition, a subgroup of patients develop severe ventricular arrhythmias that are a significant cause of sudden cardiac death in young adults. Arrhythmic MVP is defined as the presence of mitral valve prolapse with or without mitral annulus disjunction (MAD) combined with frequent ventricular ectopy, complex ectopy or sustained ventricular arrhythmia in the absence of another well-defined arrhythmic substrate. In these patients, ventricular arrhythmias most commonly originate from the mitral annulus, papillary muscles and outflow tracts. Several risk markers have been proposed, but clinical risk stratification remains challenging. Ventricular arrhythmias in patients with arrhythmic mitral valve prolapse are associated with excess long-term mortality.

There is no established medical therapy to suppress ventricular arrhythmias and relieve arrhythmic symptoms in these patients, and conventional beta-blocker therapy is often unsuccessful for both. Invasive catheter ablation can suppress ventricular arrhythmias, and thus relieve symptoms, in a subset of patients. However, many patients have multifocal ventricular ectopy, often originating from deep in the myocardium or papillary muscles and not easily accessible for catheter ablation. Furthermore, recurrence of ventricular arrhythmias is common despite initial successful catheter ablation procedures. The only strategy to prevent sudden cardiac death for high-risk patients is to implant an implantable cardioverter defibrillator (ICD), but this approach does not provide any symptomatic relief. Thus, most patients with arrhythmic mitral valve prolapse lack effective treatment options with proven efficacy in clinical trials.

Flecainide is a class 1c antiarrhythmic drug with a potent sodium channel-blocking effect frequently used in atrial tachyarrhythmias. Flecainide was developed as a treatment for ventricular arrhythmias, but its use subsided due to safety concerns when used in patients with acute myocardial infarction. However, this knowledge stems from a patient population before modern revascularization strategies after myocardial infarction and is extrapolated to patients with other structural heart diseases. Lately, flecainide has been shown to be safe in patients with stable coronary artery disease. Furthermore, flecainide reduces ventricular arrhythmias in patients with premature ventricular complex (PVC)-mediated cardiomyopathy, arrhythmogenic cardiomyopathy and catecholaminergic polymorphic ventricular tachycardia without short-term adverse effects. However, flecainide has not been studied in arrhythmic mitral valve prolapse patients.

The main goal of FLECAPRO is to evaluate the effect and safety of adding flecainide to standard beta-blocker therapy to reduce the burden of ventricular arrhythmias in patients with arrhythmic mitral valve prolapse. We hypothesize that a flecainide-based strategy is superior to a beta blocker-based strategy to suppress ventricular arrhythmias in patients with arrhythmic mitral valve prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older at the time of signing the informed consent.
* Participants must have mitral valve prolapse evident by echocardiography or cardiac magnetic resonance imaging, defined as more than or equal to 2 mm atrial displacement of any part of the mitral leaflets.
* Participants must have ventricular arrhythmias, defined as at least one of the following (i) premature ventricular complex burden ≥3% per 24 hours by Holter monitoring, (ii) premature ventricular complex burden ≥1% per 24 hours if multifocal or occurring in bi-/trigemini and/or couplets by Holter monitoring, (iii) sustained or non-sustained ventricular tachycardia, (iv) aborted cardiac arrest.
* Participants must have a clinical indication for antiarrhythmic treatment due to ventricular arrhythmias.
* Participants must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
* Participants (only women of childbearing) must accede to mandatory use of a contraceptive method for the duration of the trial and until 3 days after discontinuation of study medication.

Exclusion Criteria:

* Strict contraindications to flecainide or metoprolol use
* Heart failure (signs or symptoms, elevated N-terminal proBNP)
* Abnormal liver or kidney function (Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) three times upper normal, estimated glomerular filtration (eGRF) <60)
* Prior myocardial infarction or ischemic heart disease
* Ion channelopathy, including Brugada syndrome and long QT syndrome
* Genetic cardiomyopathy (hypertrophic cardiomyopathy, arrhythmogenic cardiomyopathy, dilated cardiomyopathy, including genotype positive phenotype negative individuals)
* Atrial flutter or permanent atrial fibrillation
* Sinus node dysfunction
* Ongoing electrolyte disorders
* More than moderate valvular disease according to international guidelines
* Pre-excitation
* Any degree of AV-block, except due to enhanced vagal tone (e.g. Wenckebach-block at night in young athletes or 1st-degree AV block that disappears during exercise)
* Bundle branch block (QRS duration >120 ms) or intraventricular conduction defect with QRS >120 ms.
* Prior flecainide therapy.
* Concomitant use of the following medications (i) CYP2D6 inhibitors/inducers, (ii) class I, III or IV antiarrhythmic drugs, (iii) clozapine, quinidine, cimetidine, bupropion, or (iii) monoamineoxidase (MAO) inhibitors
* Pregnancy
* Not willing to use a mandatory contraceptive method for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of ventricular tachyarrhythmias | 12 months
  Sum of ventricular fibrillation and ventricular tachycardia (broad complex tachycardia with heart rate >140/min) on implantable loop recorder during 12 months. Intention-to-treat, superiority.

SECONDARY OUTCOMES:
Burden of premature ventricular complexes | 12 months
  First hierarchical key secondary outcome. Assessed by 24-hour Holter monitoring. Intention-to-treat, superiority
Change in health-related quality of life | 12 months
  Second hierarchical key secondary outcome. Number of patients with ≥5-point increase in Short Form 36 overall summary score. Intention-to-treat, superiority
Number of severe ventricular tachycardias | 12 months
  Third hierarchical key secondary outcome. Sum of (i) non-sustained ventricular tachycardia with syncope, (ii) sustained ventricular tachycardia and (iii) ventricular fibrillation. Intention-to-treat, superiority
Safety composite | 12 months
  Sum of (i) number of adverse events, (ii) number of serious adverse events, and (iii) higher degree atrioventricular (AV)-block (Mobitz type 2 or 3rd-degree AV-block). Safety population.

OTHER OUTCOMES:
Number of ventricular tachycardias | 12 months
  Exploratory outcome of the individual component of the primary endpoint. Ventricular tachycardia (broad complex tachycardia with heart rate >140/min) on implantable loop recorder during 12 months.
Number of ventricular fibrillations | 12 months
  Exploratory outcome of the individual component of the primary endpoint. Ventricular fibrillations on implantable loop recorder during 12 months.
Burden of premature ventricular complexes | 12 months
  Exploratory outcome of the individual component of key secondary endpoints. Assessed by 24-hour Holter monitoring
Health-related quality of life | 12 months
  Exploratory outcome of the individual component of key secondary endpoints. Number of patients with ≥5-point increase in Short Form 36 overall summary score.
Number of severe ventricular arrhythmias | 12 months
  Exploratory outcome of the individual component of key secondary endpoints. Sum of (i) non-sustained ventricular tachycardia with syncope, (ii) sustained ventricular tachycardia and (iii) ventricular fibrillation.
Cardiac function | 12 months
  Exploratory outcome. Change in left ventricular ejection fraction assessed by echocardiography.
N-terminal pro-B-type natriuretic peptide | 12 months
  Exploratory outcome. Assessment of blood samples.
Change in New York Heart Association (NYHA) class | 12 months
  Exploratory outcome.
Change in T-wave inversions | 12 months
  Exploratory outcome. Assessed by 12-lead ECG
Change in degree of mitral regurgitation | 12 months
  Exploratory outcome. Assessed by echocardiography.
Change in health-related quality of life - Hospital Anxiety and Depression Scale questionnaire | 12 months
  Exploratory outcome. Assessed by change in the Hospital Anxiety and Depression Scale (HADS) questionnaire (0-21 with higher scores indicating greater anxiety or depression).
Primary endpoint sensitivity analysis | 12 months
  Exploratory outcome. Sum of ventricular fibrillation and ventricular tachycardia (broad complex tachycardia with heart rate >140/min) on implantable loop recorder during 12 months. Per-protocol sensitivity analysis.
Secondary safety endpoint sensitivity analysis | 12 months
  Exploratory outcome. Sum of (i) number of adverse events, (ii) number of serious adverse events, and (iii) higher degree AV-block (Mobitz type 2 or 3rd-degree AV-block). Intention-to-treat.

CONTACTS AND LOCATIONS:
Overall Officials: Eivind W Aabel, MD PhD, Principal Investigator — Department of Cardiology, Oslo University Hospital Rikshospitalet, Oslo, Norway
Locations (1):
- Oslo University Hospital Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
We will share anonymized data sets with the medical community via the medical journal upon submitting the manuscript.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be made available with the publication of the primary analysis and remain available for 1 year. Thereafter, it can be made available upon request.
Access Criteria: Researchers and clinicians with valid medical questions to be addressed. The data will not be available for commercial use.
URL: https://euclinicaltrials.eu/view-clinical-trial?p_p_id=emactview_WAR_emactpublicportlet&p_p_lifecycle=0&p_p_col_id=column-1&p_p_col_count=1&number=2022-500814-24-00

REFERENCES:
- See also: European Union Clinical Trial Information System (CTIS) application — https://euclinicaltrials.eu/view-clinical-trial?p_p_id=emactview_WAR_emactpublicportlet&p_p_lifecycle=0&p_p_col_id=column-1&p_p_col_count=1&number=2022-500814-24-00

DOCUMENTS (1):
  • Study Protocol (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT05631730/Prot_002.pdf